CLINICAL TRIAL: NCT04543903
Title: A Feasibility of Neoadjuvant Interstitial Brachytherapy (Ibt) Using Diffusing Alpha Emitters Radiation Therapy (Dart) Seeds in Men With Prostate Cancer
Brief Title: Neoadjuvant Interstitial Brachytherapy Using Diffusing Alpha Emitters Radiation Therapy in Men With Prostate Cancer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Alpha Tau Medical LTD. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CTP-PRST-02
Record Dates: First submitted 2020-08-30; First posted 2020-09-10 (Actual); Last update posted 2025-12-02 (Actual); Status verified 2024-11

CONDITIONS: Prostate Adenocarcinoma
Keywords: Prostate adenocarcinoma; Alpha radiation; Brachytherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- DaRT Seeds (Experimental): Intratumoral Diffusing alpha-emitters Radiation Therapy (DaRT) Seeds
  Interventions: Device: Radiation: Diffusing Alpha Radiation Emitters Therapy (DaRT)

INTERVENTIONS:
Device: Radiation: Diffusing Alpha Radiation Emitters Therapy (DaRT) — An intratumoral insertion of a seed(s), loaded with Radium-224, securely fixed in the seeds. The seeds release by recoil into the tumor short-lived alpha-emitting atoms.

SUMMARY:
A unique approach for cancer treatment employing intratumoral diffusing alpha radiation emitter device as a neo-adjuvant therapy in men with prostate cancer

DETAILED DESCRIPTION:
The study is planned as a prospective, open-label, one arm, single center trial, designed to assess the feasibility and safety of intratumoral DaRT seeds implantation for the treatment of local prostate cancer prior to surgery.

This approach combines the advantages of local intratumoral irradiation of the tumor, as used in conventional brachytherapy, with the power of the alpha radiation emitting atoms, that will be introduced in quantities considerably lower than radiation therapy already used in patients.

Prostate lesions with histopathological confirmation of adenocarcinoma will be treated using DaRT seeds in a neo-adjuvant setting.

Feasibility will be assessed by the successful delivery of DaRT seeds into the intratumoral environment. In addition, objective response rate will be assessed both by imaging and pathology.

ELIGIBILITY:
Inclusion Criteria:

* Pathologically confirmed, previously untreated, resectable prostate adenocarcinoma
* Ability to provide tissue sample from the target or its vicinity, either from an archive or undergo another biopsy to provide a fresh sample
* Medically fit for surgery
* Targetable lesion must be technically amenable for complete coverage (including 3-5mm margins) by the DaRT seeds
* Targetable lesion by either PSMA PET-CT according to PERCIST v1.0 OR by multiparametric MRI according RECIST v1.1
* Patients must be willing to undergo imaging before and after treatment with DaRT (prior to surgery)
* Lesion size ≤ 3 cm in the longest diameter
* Age ≥ 18 years old
* ECOG Performance Status Scale ≤ 1
* Subjects' life expectancy is more than 6 months
* WBC ≥ 3500/μl, granulocyte ≥ 1500/μl
* Platelet count ≥ 100,000/μl
* Calculated or measured creatinine clearance ≥ 60 cc/min
* AST and ALT ≤ 2.5 X ULN
* INR <1.4 for patients not on Warfarin
* Subjects are willing and able to sign an informed consent form

Exclusion Criteria:

* Documented evidence of distant metastases
* Prior TURP or prostate surgery
* Prior pelvic radiation
* Any prior pelvic malignancy or other malignancy in the last 5 years, except for cured non-melanoma skin cancer
* Inability to undergo MRI (i.e. permanent implanted device incompatible with MRI)
* Known hypersensitivity to any of the components of the treatment.
* Clinically significant cardiovascular disease, e.g. cardiac failure of New York Heart Association classes III-IV, uncontrolled coronary artery disease, cardiomyopathy, uncontrolled arrhythmia, uncontrolled hypertension, or history of myocardial infarction in the last 12 months.
* Any medical or psychiatric illness which in the opinion of the investigator would compromise the patient's ability to tolerate this treatment or interfere with the study endpoints.
* Patients must agree to use adequate contraception (vasectomy or barrier method of birth control) prior to study entry, for the duration of study participation and for 3 months after DaRT implant procedure
* Volunteers participating in another interventional study in the past 30 days which might conflict with the endpoints of this study or the evaluation of response or toxicity of DaRT.
* High probability of protocol non-compliance (in opinion of investigator)
* Subjects not willing to sign an informed consent

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2022-05-16 (Actual); Primary Completion 2025-10-01 (Actual); Study Completion 2025-10-01 (Actual)

PRIMARY OUTCOMES:
Feasibility of intratumoral DaRT seeds implantation | Study visit 'Day 0'
  To evaluate the feasibility of intratumoral insertion of DaRT seeds into prostate adenocarcinoma in the neoadjuvant setting. Feasibility will defined as the successful delivery of DaRT.
Safety of intratumoral DaRT seeds implantation | Study visit 'Day 0'
  To evaluate the safety of intratumoral insertion of DaRT seeds into prostate adenocarcinoma in the neoadjuvant setting.
  To evaluate the safety of intratumoral insertion of DaRT seeds into prostate adenocarcinoma in the neoadjuvant setting by the frequency and severity of acute adverse events related to DaRT. Adverse events will be assessed and graded according to Common Terminology and Criteria for adverse events (CTCAE) version 5.0.

SECONDARY OUTCOMES:
Pathological ORR | Week 4-6
  To asses the percentage of patients whose cancer shrinks or disappears after treatment using a biopsy from removed prostate.
Radiological ORR | 1 Week prior to surgery
  Radiological response rate according to PSMA-PET/ multiparametric MRI (SUV change/T2 weighting) through comparison with baseline imaging as assessed by RECIST or PERCIST.
Change in quality of life | Screening. Day 22.
  Change in disease related QoL using the EPIC questionnaires from baseline to prior to surgery
Change in quality of life | Screening. Day 22.
  Change in disease related QoL using the IPSS questionnaires from baseline to prior to surgery

OTHER OUTCOMES:
Assess DNA damage and repair | Day 40 - 60
  Assess DNA damage and repair (biomarker analysis: γH2AX foci, TUNEL, RAD51, RAD50, BRCA1, XRCC2, XRCC6) from baseline to surgery following DaRT seeds insertion.
Assess immune infiltration | Day 40 - 60
  Assess immune cell infiltration (biomarker analysis: CD34, TILs) from baseline to surgery following DaRT seeds insertion.
Biochemical response evaluation | Day 19-25, Day 68-82
  Biochemical response evaluation based on PSA levels

CONTACTS AND LOCATIONS:
Overall Officials: Tomer Charas, M.D, Principal Investigator — Radiotherapy unit at Rambam Health Care Campus, Israel
Locations (3):
- Israel (3):
  - RAMBAM Health Care Campus, Haifa
  - Carmel Medical Center, Haifa
  - Tel Aviv Medical Center, Tel Aviv

IPD SHARING:
Plan to Share IPD: No